CLINICAL TRIAL: NCT07282587
Title: A Phase 2 Study of ONC206 in Advanced Pheochromocytoma and Paraganglioma
Brief Title: Study of ONC206 (JZP3507) in Advanced Pheochromocytoma and Paraganglioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC206-002
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Pheochromocytoma and Paraganglioma; PCPG
Keywords: PCPG; ONC206; JZP3507
MeSH Terms: conditions — Paraganglioma | interventions — ONC206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Stage 1 Participants (Experimental): 150 mg ONC206 BID TIW
  Interventions: Drug: ONC206
- Stage 2: Dose 1 (Experimental): Participants receiving ONC206 at dose (To be Determined [TBD] post stage 1).
  Interventions: Drug: ONC206: Dose 1
- Stage 2: Dose 2 (Experimental): Participants receiving ONC206 at dose (TBD post stage 1).
  Interventions: Drug: ONC206: Dose 2

INTERVENTIONS:
Drug: ONC206 — 150 mg BID TIW
  Arms: Stage 1 Participants
Drug: ONC206: Dose 1
  Arms: Stage 2: Dose 1
Drug: ONC206: Dose 2
  Arms: Stage 2: Dose 2

SUMMARY:
This is a two-stage Phase 2 trial evaluating the efficacy and safety of ONC206 in participants with Pheochromocytoma and Paraganglioma (PCPG).

DETAILED DESCRIPTION:
Two-Stage Study to evaluate ONC206 as monotherapy doses:

Stage 1: Participants will receive 150mg ONC206 twice daily, on three consecutive days per week (BID TIW) in each 28-day cycle.

* Part A: Initial number of participants will be monitored.
* Part B: If a set number of participants have a response, then more participants will be enrolled and treated.

Stage 2: If Stage 1 meets the planned response, the study will proceed, and participants will be randomized 1:1 to receive 1 of 2 ONC206 dose levels.

ELIGIBILITY:
Inclusion criteria:

1. Has histologically confirmed pheochromocytoma or paraganglioma that is unresectable as determined by the Investigator.
2. Has failed, is not a candidate for, or has declined standard of care treatment for PCPG. There is no limit on the number of prior systemic therapies.
3. Must have measurable disease per RECIST v1.1, as assessed by the Investigator.
4. Has adequately controlled blood pressure defined as blood pressure ≤150/90 mmHg and with no change in antihypertensive medications (for participants with concomitant hypertension) for at least 14 days before the first dose of study treatment.
5. Is ≥18 years of age.
6. Is able to swallow oral tablets.
7. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2, assessed within 7 days before the first dose of study treatment.
8. Has laboratory test results meeting the following parameters within 14 days before the first dose of study treatment
9. Has an expected survival of at least 12 weeks, as predicted by the physician.
10. Has pharmacologic control of catecholamine-associated symptoms if participant has functional disease.

Exclusion criteria:

1. Has known hypersensitivity to ONC206 or any excipient used in the ONC206 study treatment formulation.
2. Has active cardiac disease/condition including any of the following:

   1. Corrected QT interval (QTc) >480 msec (based on the mean from triplicate electrocardiogram [ECGs] performed during Screening).
   2. History of documented congestive heart failure (New York Heart Association function classification III-IV).
   3. Unstable angina, acute myocardial infarction, or arterial bypass or percutaneous transluminal coronary angioplasty within 6 months before the first dose of study treatment.
3. Has previous exposure to ONC206 or dordaviprone (ONC201) from any source.
4. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Exceptions include participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, or Von Hippel-Lindau disease-associated tumors that do not require immediate surgery or intervention.
5. Has received any of the following interventions within the specified time periods before the first dose of study treatment or plans to receive any of the following interventions during study participation:

   * a. Any prior anticancer therapy or investigational agents within 4 weeks or 5 half-lives, whichever is shorter. Note: Denosumab and zoledronic acid are permissible.

     **i. Any treatment with somatostatin analog or lanreotide within 21 days before the baseline Positron Emission Tomography (PET) scan.
   * b. Strong cytochrome P450 (CYP) inhibitors within 14 days. c. Strong CYP inducers within 14 days. d. Any radiotherapy within 14 days. e. Any major surgery, open biopsy or significant traumatic injury within 1 month (30 days).
6. Is pregnant, breastfeeding, or planning to become pregnant while receiving study treatment or within 3 months after the last dose.
7. Has uncontrolled intercurrent illness or any other medical, psychiatric, or social condition that, in the opinion of the Investigator, may interfere with participant safety or the ability to comply with study requirements.
8. Has unresolved toxicities from previous locoregional, systemic, or any other therapies, defined as toxicities (other than Grade ≤2 neuropathy or alopecia) not yet resolved to the National Cancer Institute Common Terminology Criteria for Adverse Events Grade ≤1, or baseline and considered clinically significant; consult with Medical Monitor.
9. Has an active infection that requires systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 36 months.
  ORR defined as the number of participants with a confirmed complete response (CR) or partial response during the study, as per RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 36 months.
Time to Response (TTR) | Up to 36 months.
Disease Control Rate (DCR) | Up to 36 months.
Progression Free Survival (PFS) by RECIST v1.1 | Up to 36 months.
Overall Survival (OS) | Up to 36 months.
Change from Baseline in Antihypertensive Medication Dose | Up to 36 months.
Change from Baseline in Biochemical Response (Metanephrines/Disease Markers) | Up to 36 months.
Incidence of Adverse Events (AEs) | Up to 36 months.
Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Up to 36 months.
Number of Participants with Grade 4+ Clinical Laboratory Parameters | Up to 36 months.
Number of Participants with Clinically Significant Changes from Baseline in Electrocardiogram (ECG) Parameters | Up to 36 months.
Maximum Observed Concentration of ONC206 | Up to 36 months.
Time of Maximum Observed Concentration (Tmax) of ONC206 | Up to 36 months.
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUCinf) | Up to 36 months.
Area Under the Concentration Time Curve Over the Dosing Interval | Up to 36 months.
Terminal Half-Life (t1/2) of ONC206 | Up to 36 months.
Change from Baseline in European Organization for the Research and Treatment of Cancer Quality of Life-Core Questionnaire (EORTC-QLQ-C30) | Up to 36 months.
Change from Baseline in Functional Assessment of Cancer Therapy - Bone Pain (FACT-BP) | Up to 36 months.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UCLA, Los Angeles, California
  - Stanford, Palo Alto, California
  - U of Colorado, Aurora, Colorado
  - Miami Cancer Institute, Miami, Florida
  - U of Michigan, Ann Arbor, Michigan
  - Mayo-Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - PENN, Philadelphia, Pennsylvania
  - UTAH, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing/